CLINICAL TRIAL: NCT00295425
Title: Open, Multicenter, Randomized Clinical Trial in Patients With Moderate-Severe Psoriasis (PASI > 10) to Compare the Efficacy of Mycophenolate Mofetil Versus Cyclosporine A.
Brief Title: CYA Versus MMF for Treatment of Moderate-Severe Psoriasis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TALSB002; 4016406
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2006-10

CONDITIONS: Psoriasis
Keywords: psoriasis; randomized clinical trial; cyclosporine A; mycophenolate mofetil; immunosuppression
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: Cyclosporine A versus mycophenolate mofetil for psoriasis

SUMMARY:
Psoriasis is an immuno-mediated skin disorder, which affects about 2-3% of the population worldwide. For moderate-severe forms of psoriasis systemic immunosuppression is the treatment of choice. This clinical trial was initiated to compare the safety and effectiveness of mycophenolate mofetil and cyclosporine A for the treatment of psoriasis. Patients are randomized to receive either 2.5 mg/kg BW cyclosporine A or 1 g bid mycophenolate mofetil. If after six weeks no decrease in the PASI score occures cyclosporine A doses are increased to 5 mg/kg BW for additional six weeks. In the other arm mycophenolate mofetil is increased to 1 g tid for additional six weeks.

DETAILED DESCRIPTION:
Not needed.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe psoriasis (PASI Score equal and greated 10)
* written informed consent
* for female patients effective birth control

Exclusion Criteria:

* psoriasis arthritis
* psoriasis palmo-plantaris
* erythrodermic psoriasis
* drug-induced psoriasis
* pregnancy
* previous treatment with cyclosporine A or mycophenolate mofetil
* pregnancy
* reduced liver function
* high blood pressure
* reduced kidney function
* severe viral or bacterial infection
* 2 weeks before or after vaccinations
* innate or acquired immunodeficiency
* severe neurologic or psychiatric symptoms
* participation in other trials
* other reasons voiced by the treating physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2000-05; Study Completion 2006-10

PRIMARY OUTCOMES:
Comparison of the two treatment arms with regard to time until psoriasis recurrence.

SECONDARY OUTCOMES:
The treatment that leads to a 75% decrease of the initial PASI score.
The time until complete remission.
The time until partial remission has occured.
The rate of complete remission.
The rate of partial remission.
The cumulative cyclosporine A or mycophenolate mofetil doses.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Beissert, Professor, Principal Investigator — Department of Dermatology, University Hospital Muenster, Muenster, Germany
Locations (2):
- Germany (2):
  - Nicolas Hunzelmann, Cologne
  - Prof. Michael Sticherling, Leipzig